CLINICAL TRIAL: NCT04754633
Title: Comparison of Chest CT Findings Related to COVID-19 With RSNA and BSTI Guidelines: Correlation Between Radiologists
Brief Title: Comparison of Chest CT Findings Related to COVID-19 With RSNA and BSTI Guidelines
Status: Completed | Type: Observational
Sponsor: Seyhmus Kavak (Other)
Collaborators: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Sponsor-Investigator, Seyhmus Kavak, MD, Radiologist, Principal Investigator, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Organization: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Other Study IDs: 2020/588
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Infection Viral; CT Scan
Keywords: Coronavirus; Computed Thomography; PCR
MeSH Terms: conditions — COVID-19; Virus Diseases; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To present the first admission chest computed tomography (CT) findings of patients followed up with a diagnosis of COVID-19, and to compare the two classification systems by evaluating these findings according to the BSTI and RSNA guidelines.

DETAILED DESCRIPTION:
A total of 764 adult patients who were diagnosed with COVID-19 inpatient of researchers' hospital 2020 were included in this study. The findings were recorded as typical, indeterminate, and atypical by the RSNA guidelines and as classical COVID-19, possible COVID-19, indeterminate, and non-COVID-19 by the BSTI classification. The data obtained according to both classification systems were compared with each other.

ELIGIBILITY:
Inclusion Criteria:

1. Who had single negative RT-PCR
2. Non-optimal chest CT , insufficient data
3. <18 age of year
4. Thoracic trauma
5. Chest CT Negative

Exclusion Criteria:

1. RT-PCR positive and chest CT positive findings
2. At least two RT-PCR negative and chest CT positive findings
3. >18 age of year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who applied to the emergency department with the diagnosis of COVID-19 and had chest CT examination between 07.01.2020 and 07.20.2020.
Sampling Method: Probability Sample
Enrollment: 764 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Current study evaluating the success of the guidelines recommended by RSNA and BSTI in detecting COVID-19 disease | 1st week from the moment of first admission
  Kappa correlation analysis was performed between radiologists in the evaluation of chest CT findings of COVID-19 disease according to BSTI and RSNA guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlik Bilimleri Üniversitesi Training and Research Hospital, Diyarbakır, Turkey (Türkiye)